CLINICAL TRIAL: NCT02538367
Title: A Randomized, Double-blind/Open-label, Placebo/Active-controlled, Single/Multiple Dose, Parallel, Phase 1/2a Trial to Evaluate the Safety, Tolerability, PK , PD of YH12852 in Healthy Subjects and Patients With Functional Constipation
Brief Title: Phase 1/2a Trial of YH12852 in Healthy Subjects and Patients With Functional Constipation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: YH12852-102
Record Dates: First submitted 2015-08-21; First posted 2015-09-02 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Functional Constipation
MeSH Terms: interventions — prucalopride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- YH12852 IR 0.05mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 0.05mg
- YH12852 IR 0.1mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 0.1mg
- YH12852 IR 0.3mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 0.3mg
- YH12852 IR 0.5mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 0.5mg
- YH12852 IR 1mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 1mg
- YH12852 IR 2mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 2mg
- YH12852 IR 3mg (Experimental): Once daily
  Interventions: Drug: YH12852 IR 3mg
- YH12852 DR1 0.5mg (Experimental): Once daily
  Interventions: Drug: YH12852 DR1 0.5mg
- YH12852 DR1 1mg (Experimental): Once daily
  Interventions: Drug: YH12852 DR1 1mg
- YH12852 DR1 2mg (Experimental): Once daily
  Interventions: Drug: YH12852 DR1 2mg
- YH12852 DR1 4mg (Experimental): Once daily
  Interventions: Drug: YH12852 DR1 4mg
- YH12852 DR2 8mg (Experimental): Once daily
  Interventions: Drug: YH12852 DR2 8mg
- Prucalopride 2mg (Active Comparator): Once daily
  Interventions: Drug: Prucalopride 2mg
- Placebo (Placebo Comparator): Once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YH12852 IR 0.05mg
  Arms: YH12852 IR 0.05mg
Drug: YH12852 IR 0.1mg
  Arms: YH12852 IR 0.1mg
Drug: YH12852 IR 0.3mg
  Arms: YH12852 IR 0.3mg
Drug: YH12852 IR 0.5mg
  Arms: YH12852 IR 0.5mg
Drug: YH12852 IR 1mg
  Arms: YH12852 IR 1mg
Drug: YH12852 IR 2mg
  Arms: YH12852 IR 2mg
Drug: YH12852 IR 3mg
  Arms: YH12852 IR 3mg
Drug: YH12852 DR1 0.5mg
  Arms: YH12852 DR1 0.5mg
Drug: YH12852 DR1 1mg
  Arms: YH12852 DR1 1mg
Drug: YH12852 DR1 2mg
  Arms: YH12852 DR1 2mg
Drug: YH12852 DR1 4mg
  Arms: YH12852 DR1 4mg
Drug: YH12852 DR2 8mg
  Arms: YH12852 DR2 8mg
Drug: Prucalopride 2mg
  Arms: Prucalopride 2mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
A randomized, double-blind/open-label, placebo/active-controlled, single/multiple dose, parallel, phase 1/2a trial to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of YH12852 in healthy subjects and patients with functional constipation

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be willing and able to provide written informed consent.
2. BMI within the range 18 to 25 kg/m2.

Exclusion Criteria:

1. History of positive serologic evidence for infectious disease including HBsAg, anti-HCV, anti-HIV.
2. Clinically significant lab/ECG abnormalities in the opinion of the investigator.
3. WOCBP who are unwilling or unable to use an adequate contraceptive method to avoid pregnancy for the entire study. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, bilateral tubectomy, or bilateral oophorectomy) or is not postmenopausal. Post menopause is defined as amenorrhea for ≥ 12 consecutive months without another cause.

   Clinically acceptable contraceptive methods for this study: intrauterine devices (e.g., loop), physical barrier method (e.g., diaphragm, uterine cap, condom) with chemical barrier method (e.g., spermicide), sterile partner, practicing abstinence.
4. WOCBP who are willing to use hormonal methods or hormone-releasing device(e.g., mirena, implanon) for the entire study.
5. WOCBP who are pregnant or breastfeeding.
6. WOCBP with a positive pregnancy test prior to randomization.
7. Males who have not received a vasectomy must agree to use contraceptive methods defined in (a) and refrain from donating sperm throughout the study.
8. Presence of uncontrolled or severe medical illness.
9. Presence of a disease that require surgery at any time during the study.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Cmax (IR/DR multiple dose cohort and Multiple low-dose IR cohort) | Day 1 pre-dose (0 hr) ~ 24 hrs post-dose
AUC0-24 (IR/DR multiple dose cohort and Multiple low-dose IR cohort) | Day 1 pre-dose (0 hr) ~ 24 hrs post-dose
Tmax(IR/DR multiple dose cohort and Multiple low-dose IR cohort) | Day 1 pre-dose (0 hr) ~ 24 hrs post-dose
C(IR multiple dose cohort) | Day 5, 10, 12 and 13
  CD5, CD10, CD12, CD13
Cmax,ss(IR/DR multiple dose cohort and Multiple low-dose IR cohort) | Day 14
Cmax,ss (DR single dose cohort) | Day 1: pre-dose (0 hr) ~ 62hr and 86 hrs post-dose
AUClast (DR single dose cohort) | Day 1: pre-dose (0 hr) ~ 62hr and 86 hrs post-dose
C(DR multiple dose cohort and Multiple low-dose IR cohort) | Day 5, 13 and 14
  CD5, CD13, CD14

CONTACTS AND LOCATIONS:
Overall Officials: Howard Lee, MD, PhD, Principal Investigator — Department of Clinical Pharmacology and Therapeutics, Seoul National University Hospital and College of Medicine
Locations (1):
- Seoul National University Hospital, Seoul, South Korea